CLINICAL TRIAL: NCT01888549
Title: Efficacy of Proton Pump Inhibitor for Chronic Cough Caused by Gastroesophageal Reflux; Double-blind, Placebo-controlled, Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2011-0103
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Cough Caused by Gastroesophageal Reflux
Keywords: Chronic cough, proton pump inhibitor, GERD, nonacid reflux,
MeSH Terms: conditions — Chronic Cough; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- arm1-High dose PPI (Experimental)
  Interventions: Drug: High-dose PPI
- arm2-standard dose PPI (Active Comparator)
  Interventions: Drug: standard PPI
- arm3-placebo (Placebo Comparator): Esomeprazole placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: High-dose PPI — :40mg, po(per oral) 2times.day, 8weeks
  Arms: arm1-High dose PPI
Drug: standard PPI — : 40mg, po(per oral) 1times.day, 8weeks
  Arms: arm2-standard dose PPI
Drug: placebo
  Arms: arm3-placebo

SUMMARY:
Efficacy of proton pump inhibitor for chronic cough caused by gastroesophageal reflux; double-blind, placebo-controlled, randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

ages of 18 and 70 years had chronic cough of >8 weeks in duration

Exclusion Criteria:

1. abnormal chest X ray, PNS view 2. previous surgical or endoscopic antireﬂux procedure 3. previous aerodigestive malignancy or Barrett's oesophagus 4. current smokers or ex-smok-ers (deﬁned as those who quit smoking <3 months prior to study enrolment or those who have quit, but have a 20 pack year smoking history) 5. Malignancy History (lung cancer, esophageal cancer etc.) 6. upper respiratory infection within 8 weeks of study enrolment 7. currently using a PPI, H2 blocker, beta-blocker, angiotensin-converting enzyme inhibitor, corticosteroid, methylxanthine, inhaled beta-agonist, anti-inﬂammatory agent or anticholinesterase drug at time of enrolment

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
change in LCQ score and cough VAS, comparing PPI-treated group to placebo | change in LCQ score after 4 weeks and 8 weeks

SECONDARY OUTCOMES:
change in LCQ score and cough VAS, comparing PPI-treated group to placebo | change in cough VAS after 4weeks and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam severance hospita, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Park HJ, Park YM, Kim JH, Lee HS, Kim HJ, Ahn CM, Byun MK. Effectiveness of proton pump inhibitor in unexplained chronic cough. PLoS One. 2017 Oct 10;12(10):e0185397. doi: 10.1371/journal.pone.0185397. eCollection 2017. PMID 29016626